CLINICAL TRIAL: NCT05351398
Title: The Clinical Efficacy of Patient-derived Organoid-based Drug Sensitive Neoadjuvant Chemotherapy Versus Traditional Neoadjuvant Chemotherapy in Advanced Gastric Cancer: a Prospective Multi-center Randomized Controlled Study
Brief Title: The Clinical Efficacy of Drug Sensitive Neoadjuvant Chemotherapy Based on Organoid Versus Traditional Neoadjuvant Chemotherapy in Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Collaborators: Ruijin Hospital (Other); Shanghai OneTar Biomedicine Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: MISC-WXXR-002
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Advanced Gastric Carcinoma
Keywords: advanced gastric carcinoma; patient-derived organoid; personalized treatment; Neoadjuvant Chemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDO group: Patients with stage III gastric cancer who need neoadjuvant chemotherapy before radical surgery are recruited. And they are treated with individualized neoadjuvant therapy under the guidance of a patient-derived organoid (PDO)-based drug sensitivity assay.
  Interventions: Drug: PDO group; Drug: Traditional group
- Traditional group: Patients with stage III gastric cancer who need neoadjuvant chemotherapy before radical surgery are recruited. In this group, patients are treated with the SOX regimen.
  Interventions: Drug: PDO group; Drug: Traditional group

INTERVENTIONS:
Drug: PDO group — Patients with stage III gastric cancer who need neoadjuvant chemotherapy before radical surgery are recruited. And they are treated with individualized neoadjuvant therapy under the guidance of a patient-derived organoid (PDO)-based drug sensitivity assay.
Drug: Traditional group — Patients with stage III gastric cancer who need neoadjuvant chemotherapy before radical surgery are recruited. In this group, patients are treated with the SOX regimen.

SUMMARY:
Neoadjuvant chemotherapy has become the mainstream recommended treatment for advanced gastric cancer. However, due to the heterogeneity of gastric cancer, part of some patients fail to benefit from the treatment. This project aims to compare the clinical efficacy of individualized neoadjuvant therapy based on patient-derived organoid drug sensitivity assay and traditional regimen, exploring the advantages and disadvantages of these two treatments. And access the safety and clinical value of the personalized neoadjuvant therapy based on patient-derived organoid drug sensitivity assay in advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* A biopsy proven histological diagnosis of gastric adenocarcinoma or high-grade intraepithelial neoplasia
* Tumor located at stomach
* Chest/abdomen/pelvis CT scans or gastric cancer staging CT scan evaluate the clinical stage of tumor as stage III:

A. preoperative staging cT3-4N1-2 B. excluding distant organ metastasis (M0)

* Eastern Cooperative Oncology Group (ECOG) score ≤1
* Willing to participate and informed consent signed

Exclusion Criteria:

* Pregnant or lactating women
* Synchronous or heterochronic malignant carcinomas
* History of malignant carcinomas
* Clinical evidence of metastasis
* Abnormal heart, lung, liver, kidney, hematopoietic function and bone marrow reserve function, unable to tolerate surgical treatment and chemotherapy
* Mental illness or other serious cardiovascular disease
* Emergency procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastric cancer whose tumor is located in the stomach and need neoadjuvant therapy before radical surgery.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | an average of 1 year
  proportion of patients whose tumor volume reduced to a predetermined value and maintain the minimum time limit.

SECONDARY OUTCOMES:
postoperative complication | an average of 1 year
  postoperative complication
postoperative tumor regression grading | an average of 1 year
  grade the pathological response of tumor after neoadjuvant treatment, which is usually classified according to the proportion of fibrosis and residual tumor in tumor tissues.
3-year recurrence rate | an average of 3 year
  proportion of patients who relapse within 3 years after operation
chemotherapy tolerance and adverse reaction rate | an average of 1 year
R0 resection rate | an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sun, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahnghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cao W, Chen HD, Yu YW, Li N, Chen WQ. Changing profiles of cancer burden worldwide and in China: a secondary analysis of the global cancer statistics 2020. Chin Med J (Engl). 2021 Mar 17;134(7):783-791. doi: 10.1097/CM9.0000000000001474. PMID 33734139
- [Result] Kanaji S, Suzuki S, Matsuda Y, Hasegawa H, Yamamoto M, Yamashita K, Oshikiri T, Matsuda T, Nakamura T, Sumi Y, Kakeji Y. Recent updates in perioperative chemotherapy and recurrence pattern of gastric cancer. Ann Gastroenterol Surg. 2018 Aug 29;2(6):400-405. doi: 10.1002/ags3.12199. eCollection 2018 Nov. PMID 30460342
- [Result] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Result] Oh SY, Kwon HC, Jeong SH, Joo YT, Lee YJ, Cho Sh, Kang MH, Go SI, Lee GW, Kim Hg, Kang JH. A phase II study of S-1 and oxaliplatin (SOx) combination chemotherapy as a first-line therapy for patients with advanced gastric cancer. Invest New Drugs. 2012 Feb;30(1):350-6. doi: 10.1007/s10637-010-9507-2. Epub 2010 Aug 13. PMID 20706861
- [Result] Xu R, He X, Wufuli R, Su Y, Ma L, Chen R, Han Z, Wang F, Liu J. Choice of Capecitabine or S1 in Combination with Oxaliplatin based on Thymidine Phosphorylase and Dihydropyrimidine Dehydrogenase Expression Status in Patients with Advanced Gastric Cancer. J Gastric Cancer. 2019 Dec;19(4):408-416. doi: 10.5230/jgc.2019.19.e40. Epub 2019 Nov 13. PMID 31897343
- [Result] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Result] Driehuis E, Clevers H. CRISPR/Cas 9 genome editing and its applications in organoids. Am J Physiol Gastrointest Liver Physiol. 2017 Mar 1;312(3):G257-G265. doi: 10.1152/ajpgi.00410.2016. Epub 2017 Jan 26. PMID 28126704